CLINICAL TRIAL: NCT04347109
Title: cArdiac Non Invasive MApping in resynchronizaTION Registry
Brief Title: cArdiac Non Invasive MApping in resynchronizaTION
Acronym: ANIMATION
Status: Suspended | Type: Observational
Why Stopped: Organization not finalized
Sponsor: University Hospital, Tours (Other)
Responsible Party: Principal Investigator, Laurent Fauchier, Professor, University Hospital, Tours
Other Study IDs: ANIMATION Registry
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Resynchronization Therapy
Keywords: non invasive mapping; cardiac resynchronization therapy; pacing-induced cardiomyopathy; electrical shock

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biventricular Pacing: Patients implanted with a device enabling cardiac resynchronization therapy.
  Interventions: Diagnostic Test: Non invasive epicardial mapping
- Right Ventricular Pacing: Patients implanted with a right ventricular pacing device.
  Interventions: Diagnostic Test: Non invasive epicardial mapping

INTERVENTIONS:
Diagnostic Test: Non invasive epicardial mapping — Non invasive mapping using Cardio Insight system is performed in all included patients.
  Other Names: Cardio Insight system; ECG imaging

SUMMARY:
Non-invasive mapping using the Cardio Insight system is performed in heart failure patients requiring biventricular pacing to optimize therapy, and understand mechanisms underlying pacing-induced cardiomyopathy and ventricular arrhythmias.

DETAILED DESCRIPTION:
Non-invasive mapping using the Cardio Insight system is prospectively performed routinely in heart failure patients requiring cardiac resynchronization therapy.

Control patients are included, requiring chronic permanent right ventricular pacing.

Specific focus include: optimization of programming parameters, pacing-induced cardiomyopathy, ventricular arrhythmias, defibrillation threshold testing and electrical shocks.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with a biventricular pacing device (CRT) device
* Patients chronically implanted with a right ventricular pacing device.

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients referred for change or upgrading of a right ventricular pacing device in our center (CHU Tours).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ventricular activation map | Up to 6 months
  Differences (qualitative and quantitative measurements) in ventricular activation patterns are identified.
Response to CRT | Up to 2 years
  Composite endpoint : volumetric response, heart failure hospitalizations, and all-cause mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Tours, Tours, Please Select..., France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Upon submission to a peer-reviewed journal.